CLINICAL TRIAL: NCT06890546
Title: Effect of Nigella Sativa Oil Supplementation and Dietary Intervention on Lipid Profile in Overweight Adults with Hyperlipidemia: a Randomized Controlled Clinical Trial
Brief Title: Nigella Sativa Supplementation in Hyperlipidemia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Head of Nutrition and Dietetics Department, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSHYPERLIPIDEMIA
Record Dates: First submitted 2025-03-09; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hyperlipidaemia; Hyperlipidemia
Keywords: Nigella sativa; Obesity; medical nutrition therapy
MeSH Terms: conditions — Hyperlipidemias; Obesity | interventions — Nigella sativa oil; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nigella Sativa Group (Experimental): Nigella Sativa oil supplement and low calorie diet intervention
  Interventions: Dietary Supplement: Nigella Sativa Oil capsule; Behavioral: Diet
- Control Group (Placebo Comparator): low calorie diet intervention
  Interventions: Behavioral: Diet

INTERVENTIONS:
Dietary Supplement: Nigella Sativa Oil capsule — 8 weeks 2 x 900 mg Nigella Sativa oil capsule daily
  Arms: Nigella Sativa Group
Behavioral: Diet — Low calorie diet intervention

SUMMARY:
Hyperlipidemia is defined as an elevation of plasma cholesterol, lipid, or lipoprotein levels above normal due to abnormal fat metabolism or function, and individuals with hyperlipidemia are approximately twice as likely to develop cardiovascular disease. The first approach to treating hyperlipidemia is lifestyle changes, including dietary therapy and physical activity. In addition to traditional methods, treatments also include pharmacological interventions, and research on natural products and complementary therapies is increasing to increase the effectiveness of these treatment approaches. In this context, Nigella Sativa (NS) oil has emerged as a promising natural option in the treatment of hyperlipidemia and obesity in recent years.

The aim of this study was to examine the effects of NS oil supplementation given together with dietary intervention in individuals diagnosed with mild obesity.

The main questions it aims to answer are:

* Does Nigella Sativa supplementation improve blood lipid profiles in overweight or obese individuals?
* Does Nigella Sativa supplementation improve body composition in overweight or obese individuals?

Participants were individuals who were diagnosed with hyperlipidemia according to American Heart Association criteria as a result of medical evaluation by a cardiologist and who were deemed appropriate to use black seed oil supplements. Those who volunteered to participate in the study were included in the study.

The researchers are examining whether there is any effect on biochemical and anthropometric parameters by giving Nigella Sativa supplementation to a group in addition to a low-calorie diet for eight weeks.

DETAILED DESCRIPTION:
This research, which is a randomized controlled intervention study, was conducted between June 2023 and February 2024 with adult individuals with a BMI>25 kg/m2 who applied to the Cardiology Polyclinic of Karamürsel State Hospital and were referred to a nutrition and diet specialist after being diagnosed with hyperlipidemia according to AHA criteria by the physician.

Sample Selection and Randomization The sample size of the study was calculated using the G-Power 3.1.9 analysis program with a medium effect size (d=0.60), 90% power, α: 0.05 and 1-β: 0.95, with a minimum of 32 people in each group, 64 people were included. The 64 people who met the inclusion criteria were assigned to the intervention (n=32) and control (n=32) groups using the block randomization method, with similar age and gender.

Inclusion Criteria from the Study Individuals who were diagnosed with hyperlipidemia between the ages of 18-65, who did not have any serious comorbidities (kidney, liver and immune deficiency, oncological and psychiatric diseases), who were not pregnant or breastfeeding, who did not take any nutritional supplements including black seed, who did not have a known history of allergy to black seed and its products, who did not use medications that could interact with black seed oil (anticoagulant, antihypertensive, etc.), who did not use antilipidemic or anticholesterolemic medications, who did not do heavy exercise, who did not consume alcohol regularly and who did not have any special diet requirements were included in the study.

Data Collection Tools Research data were recorded using a questionnaire form, anthropometric measurements, biochemical tests and the IPAQ form.

Survey Form: Sociodemographic information, smoking and nutritional habits of the participants were recorded in the survey form.

Anthropometric Measurements: At the beginning and end of the study, body weights and analyses were performed using a bioelectrical impedance (BIA) device (Tanita Perfecto) with a sensitivity of 50 grams in accordance with the measurement standards. According to the BIA analysis, fat ratio (%), fat mass, fat-free mass, muscle mass and total body water were evaluated. At the beginning and end of the study, waist, hip and neck circumferences were measured with a non-stretchable tape measure, paying attention to anthropometric measurement standards. Waist/height and waist/hip values were calculated. Height (cm) was measured with a stadiometer in the Frankfort plane, standing and with the head upright. The body mass index (BMI) of the participants was calculated according to the body weight (kg) / height (m)2 formula and classified according to the World Health Organization (WHO) criteria.

International Physical Activity Questionnaire Short Form (IPAQ): IPAQ-Short form, developed by Craig et al. and whose Turkish validity and reliability study was conducted by Öztürk, was used to assess the physical activity levels of the participants. Physical activity levels were classified as light, moderate and vigorous active.

Biochemical Tests: Participants' biochemical tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, fasting blood glucose, ALT and AST) were analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.

Research Plan In this study, 64 hyperlipidemic individuals with BMI>25 kg/m2 were divided into 2 groups as control (n=32 individuals) and intervention (n=32 individuals). The control group was given a low-fat, low-cholesterol weight loss diet specific to the individual for 8 weeks, while the intervention group (n=32) was given a similar diet along with 2x900 mg black seed oil in softgels. Questions regarding the participants' sociodemographic characteristics, smoking, alcohol consumption and physical activity habits were recorded on a questionnaire form through face-to-face interviews. Participants attended face-to-face dietician control interviews every two weeks to observe compliance with the nutrition programs throughout the study.

Diet Plan: While determining the daily energy needs of the participants, the resting metabolic rate was calculated with the Mifflin-St.Jeor formula. The physical activity levels of the individuals were determined using the IPAQ-Short Form. The thermic effect of the nutrients was taken as 10% and the total daily energy requirement was calculated. In order for the participants to lose weight, 500 calories were subtracted from the total energy requirement. A nutrition program was given in accordance with the diet recommendations created by the American Heart Association (AHA) for hyperlipidemic individuals.

Black seed oil: In this study, black seed oil in the form of 900 mg softgels was administered orally to the intervention group at a dose of 2x900 mg. Black seed oil obtained by the cold-pressing method (TAB İlaç Sanayi A.Ş., Esenyurt, İstanbul) is in softgel form. The product is a licensed supplement with the TR-34-K-210340 certificate by the Turkish Standards Institute (TSE) and the Food Supplement Approval Number 003683-21.12.2017 of the Ministry of Agriculture and Forestry. Some studies investigating the effects of black seed oil on hyperlipidemia and other health problems show that 1-2 g of black seed or 500-1000 mg of black seed oil per day may be effective. These doses are usually taken in two divided doses daily. Moreover, a daily therapeutic dose of 2000 mg N.S has been considered safe in previous studies. Human and animal models showed no serious side effects or toxicological effects caused by the plant. The black seed oil capsules given to the participants were provided by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Adults individuals who were diagnosed hyperlipidemia
* Individuals suitable for taking Nigella satvia supplement
* Individuals BMI>25 kg/m2

Exclusion Criteria:

* Chronic liver disease,
* Chronic kidney disease,
* Heart failure, infarction or cerebrovascular disease,
* Pregnant and breastfeeding women,
* Severe psychiatric disorders,
* Oncological diseases,
* Individuals using medications that could interact with black seed oil (anticoagulant, antihypertensive, etc.)
* Individuals using antilipidemic or anticholesterolemic medications
* Individuals did not do heavy exercise
* Individuals using any nutritional supplement
* Individuals have a known history of allergy
* Individuals did not consume alcohol regularly
* Individuals with special dietary needs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Biochemical Measurements - fasting blood glucose | 8 weeks
  fasting blood glucose (mg/dL) were analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse
Biochemical Measurement | 8 weeks
  Participants' biochemical tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, (mg/dL) were analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - Liver Enzymes | 8 weeks
  Participants' liver enzymes tests (ALT and AST) (IU) were analyzed in the hospital biochemistry laboratory using routine methods at the beginning and end of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Anthropometric Measurements - Body weight (kg) | 8 weeks
  At the beginning and end of the study, body weights (kg) were measured using a bioelectrical impedance (BIA) device (Tanita Perfecto) with a sensitivity of 50 grams in accordance with the measurement standards.
Anthropometric Measurements - Height | 8 weeks
  Height (cm) was measured with a stadiometer in the Frankfort plane, standing and with the head upright.
Body Mass Index | 8 weeks
  The body mass index (BMI) of the participants was calculated according to the body weight (kg) / height (m)2 formula.
Body Mass Index Classification | 8 weeks
  The body mass index (BMI) of the participants was classified according to the World Health Organization (WHO) criteria. BMI ≥ 25 kg/m2 was overweight and ≥ 30 kg/m2 was obese.
Anthropometric Measurements - Fat Mass | 8 weeks
  Body fat mass (kg) was analyzed using a bioelectrical impedance (BIA) device (Tanita Perfecto) at the beginning and end of the study, paying attention to measurement standards.
Anthropometric Measurements - Fat ratio calculation | 8 weeks
  At the beginning and end of the study, body composition analyses were performed using a bioelectrical impedance (BIA) device (Tanita Perfecto) with the measurement standards. According to the BIA analysis, fat ratio (%) was calculated as the ratio of total body fat weight to total body weight as a percentage.
Anthropometric Measurements - Fat-free mass | 8 weeks
  Fat-free mass (kg) was analyzed using a bioelectrical impedance (BIA) device (Tanita Perfecto) at the beginning and end of the study, paying attention to measurement standards.
Anthropometric Measurements - Muscle mass | 8 weeks
  Muscle mass (kg) was analyzed using a bioelectrical impedance (BIA) device (Tanita Perfecto) at the beginning and end of the study, paying attention to measurement standards.
Anthropometric Measurements - Total body water | 8 weeks
  Total body water (kg) was analyzed using a bioelectrical impedance (BIA) device (Tanita Perfecto) at the beginning and end of the study, paying attention to measurement standards.
Anthropometric Measurements - Waist circumference | 8 weeks
  At the beginning and end of the study, waist circumference were measured with a non-flexible tape measure at the midpoint between the lowest rib bone and the cristailiac crest.
Anthropometric Measurements - Hip circumference | 8 weeks
  At the beginning and end of the study, in measuring hip circumference, the individual was asked to stand upright with their arms at their sides and their feet side by side. Frankfort plane was provided. The individual stood on their right side. The highest point on the hip (from the side) was determined and the circumference was measured with a tape measure.
Anthropometric Measurements - Neck circumference | 8 weeks
  At the beginning and end of the study, neck circumference measurement was made with a tape measure just below the laryngeal prominence (Adam's apple).
Anthropometric Measurements - Waist/Height Ratio | 8 weeks
  At the beginning and end of the study, waist/height ratio was obtained by dividing waist circumference by height.
Anthropometric Measurements - Waist/Hip Ratio | 8 weeks
  Waist/hip ratio was obtained by dividing waist circumference by hip circumference.

SECONDARY OUTCOMES:
Physical Activity | 1 week
  International Physical Activity Questionnaire Short Form developed by Craig et al. and whose Turkish validity and reliability study was conducted by Öztürk, was used to assess the physical activity levels of the participants. Physical activity levels were classified as light, moderate and vigorous active.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Seven Avuk, PhD, Principal Investigator — İstanbul Bilgi University
Locations (1):
- İstanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adanir SS, Kervancioglu P, Bahsi I, Al Saadi M, Van de Heyning P, Topsakal V. Anatomical investigation of safety determining factors for keyhole drilling trajectories for robotic cochlear implant surgery. Eur Arch Otorhinolaryngol. 2025 Jun;282(6):3037-3050. doi: 10.1007/s00405-024-09198-4. Epub 2025 Jan 17. PMID 39825202
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Norgan NG. Laboratory and field measurements of body composition. Public Health Nutr. 2005 Oct;8(7A):1108-22. doi: 10.1079/phn2005799. PMID 16277823
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Al Asoom L. Is Nigella sativa an Effective Bodyweight Lowering Agent and a Mitigator of Obesity Risk? A Literature Review. Vasc Health Risk Manag. 2022 Jul 12;18:495-505. doi: 10.2147/VHRM.S373702. eCollection 2022. PMID 35855753
- [Background] Sahebkar A, Beccuti G, Simental-Mendia LE, Nobili V, Bo S. Nigella sativa (black seed) effects on plasma lipid concentrations in humans: A systematic review and meta-analysis of randomized placebo-controlled trials. Pharmacol Res. 2016 Apr;106:37-50. doi: 10.1016/j.phrs.2016.02.008. Epub 2016 Feb 10. PMID 26875640
- [Background] Rounagh M, Musazadeh V, Hosseininejad-Mohebati A, Falahatzadeh M, Kavyani Z, Rostami RB, Vajdi M. Effects of Nigella sativa supplementation on lipid profiles in adults: An updated systematic review and meta-analysis of randomized controlled trials. Clin Nutr ESPEN. 2024 Jun;61:168-180. doi: 10.1016/j.clnesp.2024.03.020. Epub 2024 Mar 22. PMID 38777430
- [Background] Lichtenstein AH, Appel LJ, Vadiveloo M, Hu FB, Kris-Etherton PM, Rebholz CM, Sacks FM, Thorndike AN, Van Horn L, Wylie-Rosett J. 2021 Dietary Guidance to Improve Cardiovascular Health: A Scientific Statement From the American Heart Association. Circulation. 2021 Dec 7;144(23):e472-e487. doi: 10.1161/CIR.0000000000001031. Epub 2021 Nov 2. PMID 34724806
- [Background] Karr S. Epidemiology and management of hyperlipidemia. Am J Manag Care. 2017 Jun;23(9 Suppl):S139-S148. PMID 28978219
- [Background] Kaatabi H, Bamosa AO, Lebda FM, Al Elq AH, Al-Sultan AI. Favorable impact of Nigella sativa seeds on lipid profile in type 2 diabetic patients. J Family Community Med. 2012 Sep;19(3):155-61. doi: 10.4103/2230-8229.102311. PMID 23230380
- [Background] Razmpoosh E, Safi S, Nadjarzadeh A, Fallahzadeh H, Abdollahi N, Mazaheri M, Nazari M, Salehi-Abargouei A. The effect of Nigella sativa supplementation on cardiovascular risk factors in obese and overweight women: a crossover, double-blind, placebo-controlled randomized clinical trial. Eur J Nutr. 2021 Jun;60(4):1863-1874. doi: 10.1007/s00394-020-02374-2. Epub 2020 Sep 2. PMID 32876804
- [Background] Ibrahim RM, Hamdan NS, Mahmud R, Imam MU, Saini SM, Rashid SN, Abd Ghafar SA, Latiff LA, Ismail M. A randomised controlled trial on hypolipidemic effects of Nigella Sativa seeds powder in menopausal women. J Transl Med. 2014 Mar 31;12:82. doi: 10.1186/1479-5876-12-82. PMID 24685020
- [Background] Ahmad A, Husain A, Mujeeb M, Khan SA, Najmi AK, Siddique NA, Damanhouri ZA, Anwar F. A review on therapeutic potential of Nigella sativa: A miracle herb. Asian Pac J Trop Biomed. 2013 May;3(5):337-52. doi: 10.1016/S2221-1691(13)60075-1. PMID 23646296
- [Background] Qidwai W, Hamza HB, Qureshi R, Gilani A. Effectiveness, safety, and tolerability of powdered Nigella sativa (kalonji) seed in capsules on serum lipid levels, blood sugar, blood pressure, and body weight in adults: results of a randomized, double-blind controlled trial. J Altern Complement Med. 2009 Jun;15(6):639-44. doi: 10.1089/acm.2008.0367. PMID 19500003
- [Background] Mahdavi R, Namazi N, Alizadeh M, Farajnia S. Effects of Nigella sativa oil with a low-calorie diet on cardiometabolic risk factors in obese women: a randomized controlled clinical trial. Food Funct. 2015 Jun;6(6):2041-8. doi: 10.1039/c5fo00316d. PMID 26029855
- [Background] Heshmati J, Namazi N. Effects of black seed (Nigella sativa) on metabolic parameters in diabetes mellitus: a systematic review. Complement Ther Med. 2015 Apr;23(2):275-82. doi: 10.1016/j.ctim.2015.01.013. Epub 2015 Feb 9. PMID 25847566
- [Background] Zaoui A, Cherrah Y, Alaoui K, Mahassine N, Amarouch H, Hassar M. Effects of Nigella sativa fixed oil on blood homeostasis in rat. J Ethnopharmacol. 2002 Jan;79(1):23-6. doi: 10.1016/s0378-8741(01)00342-7. PMID 11744291
- [Background] Meddah B, Ducroc R, El Abbes Faouzi M, Eto B, Mahraoui L, Benhaddou-Andaloussi A, Martineau LC, Cherrah Y, Haddad PS. Nigella sativa inhibits intestinal glucose absorption and improves glucose tolerance in rats. J Ethnopharmacol. 2009 Jan 30;121(3):419-24. doi: 10.1016/j.jep.2008.10.040. Epub 2008 Nov 17. PMID 19061948
- [Background] Datau EA, Wardhana, Surachmanto EE, Pandelaki K, Langi JA, Fias. Efficacy of Nigella sativa on serum free testosterone and metabolic disturbances in central obese male. Acta Med Indones. 2010 Jul;42(3):130-4. PMID 20724766